CLINICAL TRIAL: NCT03986515
Title: Clinical Study of SHR-1210 Plus Apatinib in Patients With Advanced Mucosal Melanoma Whose Diseases Progress After Chemotherapy
Brief Title: Apatinib Plus SHR1210 in Advanced Mucosal Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH immunotherapy003
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Mucosal Melanoma; Advanced Cancer; Apatinib; SHR-1210
MeSH Terms: interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): apatinib 250mg orally once a day until disease progression of occurrence of intolerable adverse events.
  SHR-1210 200mg every two weeks until disease progression of occurrence of intolerable adverse events.
  (the first dose of SHR-1210 is set on the 3-5 days after apatinib
  Interventions: Drug: apatinib plus SHR-1210

INTERVENTIONS:
Drug: apatinib plus SHR-1210 — apatinib 250mg qd, 3-5 days later SHR-1210 200mg q3w

SUMMARY:
There is still no effective treatment for advanced mucosal melanoma at present. The efficacy of single-agent PD-1 inhibitors is less than 20%. It is urgent to explore regimens to improve the efficacy of PD-1 inhibitors in patients with advanced mucosal melanoma. This study is performed to explore the safety and efficacy of apatinib plus SHR-1210 in patients with advanced mucosa melanoma whose diseases progress after chemotherapy.

DETAILED DESCRIPTION:
Apatinib is an oral small molecule anti-angiogenesis inhibitors. It inhibits VEGFR-2 tyrosine kinase activity, thereby blocking VEGF-induced signaling and exerting a strong inhibitory effect on tumor angiogenesis.Apatinib has shown anti-melanoma activity in retrospective study. However, the efficacy is still very low. SHR-1210 is an anti-PD-1 antibody produced by Hengrui Pharmaceutical Co., Ltd. Apatinib plus SHR-1210 has shown synergy in several malignancies. This study is conducted to explore the efficacy and safety in advanced mucosa melanoma

ELIGIBILITY:
Inclusion Criteria:

* mucosal melanoma by pathology
* expected lifespan ≥ 3 months
* ECOG 0-2
* failure after one kind of chemotherapeutic regimen
* at least one measurable lesion by RECIST 1.1
* enough organ function
* blood pressure is normal; for patients with hypertension the blood pressure should be controlled in normal by antihypertensive drugs
* no other serious diseases conflicting with this regimen
* no history of other malignancies
* pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
* informed consent from the patient

Exclusion Criteria:

* Suffering from serious infectious diseases within 4 weeks before enrollment
* requiring intermittent use of bronchodilators or medical interventions
* usage of immunosuppressants before enrollment and the dose of immunosuppressant used ≥ 10mg / day oral prednisone for more than 2 weeks
* serious allergy
* serious mental diseases
* abnormal coagulation funtion,bleeding tendency or receiving thrombolytic or anticoagulant therapy
* abdominal fistula, gastrointestinal perforation, or abdominal abscess within 4 weeks prior to enrollment
* previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, severe lung damage, etc.
* other situations evaluated by investigator unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | three months
  the proportion of patients with CR, PR, and SD in the group

SECONDARY OUTCOMES:
progression-free survival | six months
  the time frame from the first day of apatinib to the date of confirmed progressive disease or death which one occurrs first.
overall survival | eighteen months
  the time frame from the first day of apatinib to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ding, Master, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China